CLINICAL TRIAL: NCT05060237
Title: A Non-randomized, Open-label, Multicenter Study to Evaluate the Safety and Tolerability of BF-200 ALA (Ameluz®) in the Expanded Field-directed Treatment of Actinic Keratosis on the Face and Scalp With Photodynamic Therapy (PDT)
Brief Title: Study to Evaluate Safety and Tolerability of BF-200 ALA (Ameluz®) for Photodynamic Therapy in the Treatment of the Expanded Field of Actinic Keratosis on Face and Scalp
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biofrontera Bioscience GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALA-AK-CT018
Record Dates: First submitted 2021-09-07; First posted 2021-09-29 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Actinic Keratosis; Keratosis, Actinic; Keratosis
Keywords: Actinic keratosis; Photodynamic therapy; 5-aminolevulinic acid; Photosensitizing Agents; Dermatologic Agents; Precancerous condition; Skin Disease
MeSH Terms: conditions — Keratosis, Actinic; Keratosis; Precancerous Conditions; Skin Diseases | interventions — BF-200 ALA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- BF-200 ALA (Experimental): Topical application of BF-200 ALA containing 7.8% 5-ALA (5-aminolevulinic acid).
  One single photodynamic therapy (PDT).
  Interventions: Combination Product: BF-200 ALA and red light LED lamp

INTERVENTIONS:
Combination Product: BF-200 ALA and red light LED lamp — Photodynamic therapy (PDT) using BF-RhodoLED® XL (ALA-PDT, Ameluz®-PDT):
  Topical application of 3 tubes BF-200 ALA on the expanded treatment field (60 cm²), followed by red light illumination with BF-RhodoLED® XL after 3 h incubation of study medication under light-tight, occlusive dressing.

SUMMARY:
The aim of the study is to evaluate the safety and tolerability of PDT for treatment of mild to severe actinic keratosis on the face and scalp in the expanded treatment field using 3 tubes of BF-200 ALA 10% gel (Ameluz®) in conjunction with the BF-RhodoLED® XL PDT lamp.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability of subjects to provide informed consent and sign the Health Insurance Portability and Accountability Act (HIPAA) form. A study-specific informed consent and HIPAA form must be obtained in writing prior to starting any study procedures.
2. Subjects with mild to severe clinically confirmed AK lesions (according to Olsen) on the face and/or scalp. In case of severe AK lesions, a biopsy must be taken for confirmation of diagnosis. At least 8 mild to moderate AK lesions with a diameter of ≥4 mm must be present in the treatment field. The treatment field (continuous or in several patches) totaling about 60 cm2 must be located within one effective illumination area. The AK lesions should be clearly distinguishable, without restrictions on the distance between lesions. Lesions should have a minimal distance of 1 cm between the lesion margin and the border of the treatment field.
3. All sexes, ≥18 years of age.
4. Willingness and ability to comply with study procedures, particularly willingness to receive a PDT session and to undergo 2 mm punch biopsy/biopsies in case of severe AK lesion(s) at the screening visit.
5. Subjects with good general health or with clinically stable medical conditions will be permitted to be included in the study. Subjects with clinically stable medical conditions will be permitted for inclusion into the study if not using prohibited medication.
6. Willingness to stop the use of moisturizers and any other non-medical topical treatments within the treatment field at least 24 h prior to the visits.
7. Acceptance to abstain from extensive sunbathing and the use of a solarium or tanning beds during the study.
8. For female subjects with reproductive potential: Negative serum pregnancy test.
9. For female subjects with reproductive potential: Effective contraception at screening visit and throughout the study.

Exclusion Criteria:

1. Any known history of hypersensitivity to ALA, porphyrins or excipients of BF-200 ALA.
2. History of soy or peanut allergy.
3. Subjects with sunburn or other possible confounding skin conditions (e.g. wounds, irritations, bleeding or skin infections) inside or in close proximity (<10 cm distance) to the treatment field.
4. Clinically significant (CS) medical conditions making implementation of the protocol or interpretation of the study results difficult or impairing subject's safety such as:

   1. Presence of photodermatoses or porphyria
   2. Metastatic tumor or tumor with high probability of metastasis
   3. Infiltrating skin neoplasia (suspected or known)
   4. Unstable cardiovascular disease (New York Heart Association class III, IV)
   5. Unstable hematologic (including myelodysplastic syndrome), hepatic, renal, neurologic, or endocrine condition
   6. Unstable collagen-vascular condition
   7. Unstable gastrointestinal condition
   8. Immunosuppressive condition
   9. Presence of clinically significant inherited or acquired coagulation defect
5. Clinical diagnosis of atopic dermatitis, Bowen's disease, basal cell carcinoma, eczema, psoriasis, rosacea, squamous cell carcinoma, other malignant or benign tumors inside or in close proximity (<10 cm distance) to the treatment field.
6. Presence of strong artificial pigmentation (e.g. tattoos) or any other abnormality that may impact lesion assessment or light penetration in the treatment field.
7. Any physical therapy such as cryosurgery, laser therapy, electrodessication, microdermabrasion, surgical removal of lesions, curettage, or treatment with chemical peels such as trichloroacetic acid inside or in close proximity (<10 cm distance) to the treatment field within 4 weeks prior to screening.
8. Any of the topical treatments defined below within the designated periods prior to screening:

   1. Topical treatment with ALA or ALA esters (e.g. methyl aminolevulinic acid (MAL)) or an investigational drug in- and outside the treatment field within 8 weeks.
   2. Topical treatment with immunosuppressive, cytostatic or cytotoxic drugs inside or in close proximity (<10 cm distance) to the treatment field within 8 weeks.
   3. Start of topical administration of a medication with hypericin or other drugs with phototoxic or photoallergic potential inside or in close proximity (<10 cm distance) to the treatment field within 4 weeks. Subjects may, however, be eligible if such medication was applied for more than 4 weeks prior to screening without evidence of an actual phototoxic/photoallergic reaction.
9. Any use of the systemic treatments within the designated periods prior to screening:

   1. Cytostatic or cytotoxic drugs within 6 months.
   2. Immunosuppressive therapies or use of ALA or ALA esters (e.g. MAL) within 12 weeks.
   3. Drugs known to have major organ toxicity within 8 weeks or an investigational drug.
   4. Interferon or glucocorticosteroids within 6 weeks.
   5. Start of intake of medication with hypericin or systemically acting drugs with phototoxic or photoallergic potential within 8 weeks prior to screening. Subjects may, however, be eligible if such medication was taken in for more than 8 weeks prior to the screening visit without evidence of an actual phototoxic/photoallergic reaction.
10. Breast feeding women.
11. Suspicion of drug or alcohol abuse.
12. Subjects unlikely to comply with protocol, e.g. inability to return for visits, unlikely to complete the study, or inappropriate in the opinion of the investigator.
13. A member of study site staff or sponsor staff directly involved in the conduct of the protocol or a close relative thereof.
14. Simultaneous participation in another clinical study.

Dosing day exclusion criteria:

At Visit 2 (baseline, PDT-1)

Subjects with sunburn or other possibly confounding skin conditions (e.g. wounds, irritations, bleeding or skin infections) inside or in close proximity (<10 cm distance) to the treatment field.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schlesinger, MD, Principal Investigator — Clinical Research Center of the Carolinas, 1364 Ashley River Road, Charleston, SC 29407, USA
Locations (9):
- United States (9):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Alliance Dermatology & Mohs Center, Phoenix, Arizona
  - Dermatology Practice, Greenwood Village, Colorado
  - Laser and Skin Surgery Center of Indiana, Indianapolis, Indiana
  - Skin Search of Rochester, Inc, Rochester, New York
  - Rochester Dermatologic Surgery, Victor, New York
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Austin Institute for Clinical Research, Houston, Texas
  - Austin Institute for Clinical Research Inc., Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: According to protocol, 100 participants were planned to be dosed. To meet this requirement, 112 participants were enrolled, resulting in 100 participants to receive treatment.
Groups:
- BF-200 ALA: Topical application of BF-200 ALA containing 7.8% 5-ALA (5-aminolevulinic acid).
  One single photodynamic therapy (PDT).
  BF-200 ALA and red light LED lamp: Photodynamic therapy (PDT) using BF-RhodoLED® XL (ALA-PDT, Ameluz®-PDT):
  Topical application of 3 tubes BF-200 ALA on the expanded treatment field (60 cm²), followed by red light illumination with BF-RhodoLED® XL after 3 h incubation of study medication under light-tight, occlusive dressing.
Period: Overall Study
Arm/Group | BF-200 ALA
Started | 112
Treated on the Face | 40
Treated on the Scalp | 39
Treated on the Face and Scalp | 21
Completed | 100
Not Completed | 12
Not completed — Withdrawal by Subject | 4
Not completed — Screening failure | 8

BASELINE CHARACTERISTICS:
Population: Subjects with mild to severe clinically confirmed AK lesions were included. At least 8 mild to moderate AK lesions with a diameter of ≥ 4 mm had to be present in the treatment field. The treatment field (continuous or in several patches) totaling about 60 cm^2 had to be located within one effective illumination area.
Groups:
- Face (BF-200 ALA): Topical application of BF-200 ALA containing 7.8% 5-ALA (5-aminolevulinic acid).
  One single photodynamic therapy (PDT).
  BF-200 ALA and red light LED lamp: Photodynamic therapy (PDT) using BF-RhodoLED® XL (ALA-PDT, Ameluz®-PDT):
  Topical application of 3 tubes BF-200 ALA on the expanded treatment field (60 cm²) on the face, followed by red light illumination with BF-RhodoLED® XL after 3 h incubation of study medication under light-tight, occlusive dressing.
- Scalp (BF-200 ALA): Topical application of BF-200 ALA containing 7.8% 5-ALA (5-aminolevulinic acid).
  One single photodynamic therapy (PDT).
  BF-200 ALA and red light LED lamp: Photodynamic therapy (PDT) using BF-RhodoLED® XL (ALA-PDT, Ameluz®-PDT):
  Topical application of 3 tubes BF-200 ALA on the expanded treatment field (60 cm²) on the scalp, followed by red light illumination with BF-RhodoLED® XL after 3 h incubation of study medication under light-tight, occlusive dressing.
- Face and Scalp (BF-200 ALA): Topical application of BF-200 ALA containing 7.8% 5-ALA (5-aminolevulinic acid).
  One single photodynamic therapy (PDT).
  BF-200 ALA and red light LED lamp: Photodynamic therapy (PDT) using BF-RhodoLED® XL (ALA-PDT, Ameluz®-PDT):
  Topical application of 3 tubes BF-200 ALA on the expanded treatment field (60 cm²) on the face and scalp, followed by red light illumination with BF-RhodoLED® XL after 3 h incubation of study medication under light-tight, occlusive dressing.
- Total: Total of all reporting groups
Arm/Group | Face (BF-200 ALA) | Scalp (BF-200 ALA) | Face and Scalp (BF-200 ALA) | Total
Number analyzed (Participants) | 40 | 39 | 21 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (7.5) | 70.1 (6.7) | 66.5 (7.9) | 67.9 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 0 | 0 | 12
  Male | 28 | 39 | 21 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 40 | 38 | 21 | 99
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 40 | 39 | 20 | 99
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Fitzpatrick skin type [Count of Participants; unit: Participants] — Skin type was evaluated according to Fitzpatrick criteria (Fitzpatrick 1988). Skin type is often categorized according to the Fitzpatrick skin type scale, which ranges from very fair (skin type I) to very dark (skin type VI). Genetic disposition (color of eyes, hair, etc), reaction to sun exposure and tanning habits (sun bathing, artificial tanning or tanning creams) influence the skin type.
  Participants
    I-II | 31 | 20 | 14 | 65
    III-IV | 9 | 19 | 7 | 35
Number of AK lesions [Mean (Standard Deviation); unit: Number of AK lesions]
  Total | 17.6 (11.0) | 15.7 (11.3) | 16.8 (11.4) | 16.7 (11.1)
  Diameter < 4 mm | 4.3 (9.9) | 4.1 (10.1) | 1.8 (3.9) | 3.7 (9.1)
  Diameter ≥ 4 mm | 13.3 (7.9) | 11.6 (4.4) | 15.0 (11.4) | 13.0 (7.8)
Total area of AK target lesions ≥ 4 mm [Mean (Standard Deviation); unit: mm ^2] | 426.5 (269.7) | 701.8 (830.6) | 626.8 (361.0) | 575.9 (579.3)
Severity of AK target lesions ≥ 4 mm [Number; unit: Number of AK lesions] — AK lesion severity was evaluated according to the Olsen Severity Grading (Olsen et al., 1991) as follows:
  * Mild/grade 1: AK lesions present as flat, pink maculae without signs of hyperkeratosis and erythema. The lesions are slightly palpable, better felt than seen.
  * Moderate/grade 2: AK lesions present as pink to reddish papules and erythematous plaques with hyperkeratotic surface. These AK lesions are moderately thick and can be easily seen and felt.
  * Severe/grade 3: AK lesions present as very thick plaques with hyperkeratotic surface. These AK lesions are thick and/or obvious.
  Number of AK lesions
    Mild/ grade 1 | 329 | 209 | 147 | 685
    Moderate/ grade 2 | 203 | 231 | 165 | 599
    Severe/ grade 3 | 0 | 12 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Frequency and Severity of Adverse Events (AEs), Serious AEs (SAEs), and Treatment Emergent Adverse Events (TEAEs).
Description: TEAEs are defined as all AEs with onset or worsening after treatment with IMP up to Visit 5 (Final Visit). TEAEs are considered being related to IMP or medical device, if causal relationship between IMP or medical device and the TEAE is at least possible or relationship assessment is missing. If an AE occurs in different treatment areas (face, scalp, face and scalp), it is reported separately for each treatment area. Thus, some AEs are counted more than once.
Time Frame: Through study completion, on average 6 weeks
Measure: Number; unit: Number of events
Groups:
- Total (BF-200 ALA): Topical application of BF-200 ALA containing 7.8% 5-ALA (5-aminolevulinic acid).
  One single photodynamic therapy (PDT).
  BF-200 ALA and red light LED lamp: Photodynamic therapy (PDT) using BF-RhodoLED® XL (ALA-PDT, Ameluz®-PDT):
  Topical application of 3 tubes BF-200 ALA on the expanded treatment field (60 cm²) on the face and/or scalp, followed by red light illumination with BF-RhodoLED® XL after 3 h incubation of study medication under light-tight, occlusive dressing.
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
Number of events
  Any AEs | 888
  Any AEs : mild | 563
  Any AEs : moderate | 242
  Any AEs : severe | 83
  Any serious AEs | 0
  Any TEAEs | 871
  Any TEAEs : mild | 546
  Any TEAEs : moderate | 242
  Any TEAEs : severe | 83
  Any serious TEAEs | 0
  Any TEAEs leading to death | 0
  Any TEAEs related to IMP | 809
  Any TEAEs related to medical device | 782
  Any TEAEs related to IMP or medical device | 811
  Any TEAEs leading to study discontinuation | 0

2. Primary Outcome: Duration of TEAEs Including the Breakdown of Severity Category (Mild, Moderate, Severe).
Description: The duration of TEAEs related to IMP and/or medical device which occurred in at least two subjects and with complete start and stop dates was analyzed. In addition, the proportion of the duration by severity was analyzed. Duration of severity per subject and preferred term is calculated in days counting all days and all episodes of one severity category together. Calculation is done referring to all subjects with occurrence of respective preferred term. If a severity category of a preferred term does not occur in a subject, the duration of this category is set to 0. If an AE occurs in different treatment areas, it is reported separately for each treatment area (face, scalp, face and scalp). Thus, some AEs are counted more than once for the analysis.
Time Frame: From treatment day (day 1, Visit 2) up to Visit 5 (approx. 28 days post treatment)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
days
  Application site discharge : all severities | 5.50 (3.32)
  Application site discharge : mild | 5.50 (3.32)
  Application site discolouration : all severities | 11.17 (5.60)
  Application site discolouration : mild | 4.33 (4.97)
  Application site discolouration : moderate | 6.83 (8.82)
  Application site discomfort : all severities | 4.55 (2.84)
  Application site discomfort : mild | 4.55 (2.84)
  Application site dryness : all severities | 12.33 (10.02)
  Application site dryness : mild | 8.00 (12.17)
  Application site dryness : moderate | 4.33 (7.51)
  Application site erosion : all severities | 8.88 (5.07)
  Application site erosion : mild | 5.59 (4.78)
  Application site erosion : moderate | 2.81 (5.37)
  Application site erosion : severe | 0.47 (1.88)
  Application site erythema : all severities | 19.04 (12.78)
  Application site erythema : mild | 10.09 (13.60)
  Application site erythema : moderate | 7.95 (10.11)
  Application site erythema : severe | 1.00 (4.80)
  Application site exfoliation : all severities | 13.62 (9.81)
  Application site exfoliation : mild | 10.48 (8.65)
  Application site exfoliation : moderate | 2.79 (6.16)
  Application site exfoliation : severe | 0.35 (1.46)
  Application site haemorrhage : all severities | 3.33 (2.74)
  Application site haemorrhage : mild | 2.28 (2.31)
  Application site haemorrhage : moderate | 1.06 (2.65)
  Application site hyperaesthesia : all severities | 6.22 (3.27)
  Application site hyperaesthesia : mild | 3.61 (2.69)
  Application site hyperaesthesia : moderate | 2.44 (4.45)
  Application site hyperaesthesia : severe | 0.17 (0.50)
  Application site induration : all severities | 15.71 (29.67)
  Application site induration : mild | 12.41 (30.72)
  Application site induration : moderate | 3.29 (4.86)
  Application site oedema : all severities | 9.76 (4.97)
  Application site oedema : mild | 6.93 (5.80)
  Application site oedema : moderate | 2.69 (3.78)
  Application site oedema : severe | 0.15 (0.86)
  Application site pain : all severities | 8.91 (7.11)
  Application site pain : mild | 4.19 (6.17)
  Application site pain : moderate | 2.84 (4.99)
  Application site pain : severe | 1.87 (3.47)
  Application site papules : all severities | 8.50 (4.95)
  Application site papules : mild | 8.50 (4.95)
  Application site paraesthesia : all severities | 3.00 (2.39)
  Application site paraesthesia : mild | 2.13 (2.29)
  Application site paraesthesia : moderate | 0.47 (0.83)
  Application site paraesthesia : severe | 0.40 (1.55)
  Application site pruritus : all severities | 9.29 (7.30)
  Application site pruritus : mild | 8.06 (7.42)
  Application site pruritus : moderate | 1.13 (3.64)
  Application site pruritus : severe | 0.10 (0.60)
  Application site pustules : all severities | 5.67 (1.53)
  Application site pustules : mild | 3.83 (2.84)
  Application site pustules : moderate | 1.83 (1.61)
  Application site scab : all severities | 10.81 (7.42)
  Application site scab : mild | 7.53 (8.52)
  Application site scab : moderate | 3.17 (4.83)
  Application site scab : severe | 0.11 (0.79)
  Application site swelling : all severities | 6.50 (3.33)
  Application site swelling : mild | 5.83 (4.22)
  Application site swelling : moderate | 0.67 (1.63)
  Application site vesicles : all severities | 5.07 (4.08)
  Application site vesicles : mild | 4.68 (4.00)
  Application site vesicles : moderate | 0.39 (1.00)
  Application site warmth : all severities | 2.13 (1.75)
  Application site warmth : mild | 0.72 (0.97)
  Application site warmth : moderate | 0.94 (1.06)
  Application site warmth : severe | 0.47 (1.12)
  Blood pressure increased : all severities | 5.50 (2.12)
  Blood pressure increased : mild | 3.50 (4.95)
  Blood pressure increased : moderate | 2.00 (2.83)
  Chills : all severities | 1.60 (0.89)
  Chills : mild | 1.20 (0.45)
  Chills : moderate | 0.40 (0.89)
  Dry Eye : all severities | 5.00 (2.65)
  Dry Eye : mild | 5.00 (2.65)
  Fatigue : all severities | 4.50 (1.29)
  Fatigue : mild | 2.25 (2.87)
  Fatigue : moderate | 2.25 (2.63)
  Headache : all severities | 2.71 (1.79)
  Headache : mild | 2.15 (2.12)
  Headache : moderate | 0.56 (0.90)
  Nausea : all severities | 1.00 (0.00)
  Nausea : mild | 0.50 (0.71)
  Nausea : moderate | 0.50 (0.71)
  Poor quality sleep : all severities | 7.50 (0.71)
  Poor quality sleep : mild | 4.00 (5.66)
  Poor quality sleep : moderate | 3.50 (4.95)

3. Primary Outcome: Assessment of New Lesions (AK, NMSC Such as BCC, SCC or Bowens Disease, and Melanoma) if They Occur Inside the Treatment Field
Description: Assessed were newly occuring lesions of actinic keratosis (AK), non-melanoma skin cancer (NMSC) such as basal cell carcinoma (BCC), squamous cell carcinoma (SCC) or Bowens disease, and melanoma inside the treatment field. Cumulative number of lesions is reported.
Time Frame: From treatment day (day 1, Visit 2) up to Visit 5 (approx. 28 days post treatment)
Measure: Number; unit: Number of lesions
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
Number of lesions
  Any new lesions | 38
  Seborrhoeic keratosis | 1
  Actinic keratosis | 36
  Milia | 1

4. Primary Outcome: Assessment of New Lesions (AK, NMSC, and Melanoma) if They Occur Around the Treatment Field at a Distance of <10 cm
Description: as for outcome 3
Time Frame: From treatment day (day 1, Visit 2) up to Visit 5 (approx. 28 days post treatment)
Measure: Number; unit: Number of lesions
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
Number of lesions
  Any new lesions | 10
  Seborrhoeic keratosis | 1
  Squamous cell carcinoma | 1
  Actinic keratosis | 8

5. Primary Outcome: Application Site Skin Reactions During and Post PDT, Assessed by the Investigator
Description: Application site skin reaction categories: discharge, erosion, erythema, exfoliation, fissure, induration, oedema, scabbing, skin flaking, ulceration, vesicles, other; severity of AE: mild, moderate or severe
Time Frame: From treatment day (day 1, Visit 2) up to Visit 5 (approx. 28 days post treatment)
Measure: Number; unit: percentage of partcipants
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
percentage of partcipants
  Any application site skin reactions | 96.0
  Application site discharge | 4.0
  Application site discolouration | 6.0
  Application site dryness | 4.0
  Application site erosion | 16.0
  Application site erythema | 86.0
  Application site exfoliation | 87.0
  Application site fissure | 1.0
  Application site haemorrhage | 10.0
  Application site induration | 18.0
  Application site oedema | 35.0
  Application site papules | 2.0
  Application site scab | 49.0
  Application site swelling | 6.0
  Application site vesicles | 14.0
  Application site pustules | 3.0

6. Primary Outcome: Application Site Discomfort During and Post PDT, Reported by the Subjects
Description: Application site discomfort categories: burning, hyperaesthesia, pain, paraesthesia, pruritus, stinging, warmth, other; severity of AE: mild, moderate or severe
Time Frame: From treatment day (day 1, Visit 2) up to Visit 5 (approx. 28 days post treatment)
Measure: Number; unit: percentage of participants
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
percentage of participants
  Any application site discomfort | 97.0
  Application site discomfort | 11.0
  Application site hyperaesthesia | 10.0
  Application site hypoaesthesia | 1.0
  Application site pain | 96.0
  Application site paraesthesia | 15.0
  Application site photosensitivity reaction | 1.0
  Application site pruritus | 65.0
  Application site warmth | 17.0

7. Primary Outcome: Application Site Pain During Illumination
Description: Assessed by the subjects using an 11-point numeric rating scale (NRS), where a score of 0 means "no pain" and a score of 10 means "worst imaginable pain".
Time Frame: At treatment day (day 1, Visit 2) after end of illumination
Population: For this study, concomitant medication as pain-relieving measure prior to illumination, concomitant medications given as pain-relieving measures during illumination and physical pain-relieving measures (i.e. interruption of the illumination and/or cooling with an air stream and/or nebulized water) were allowed. Subjects might have received a combination of medications (prior and/or during) and/or measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
score on a scale
  Overall | 7.4 (2.1)
  Without concomitant pain relieving medication prior to illumination: number analyzed (Participants) | 52
  Without concomitant pain relieving medication prior to illumination | 7.6 (1.8)
  With concomitant pain relieving medication prior to illumination: number analyzed (Participants) | 48
  With concomitant pain relieving medication prior to illumination | 7.2 (2.5)
  Without concomitant pain relieving medication during illumination: number analyzed (Participants) | 86
  Without concomitant pain relieving medication during illumination | 7.3 (2.1)
  With concomitant pain relieving medication during illumination: number analyzed (Participants) | 14
  With concomitant pain relieving medication during illumination | 8.4 (1.9)
  Without physical pain relieving measures during illumination: number analyzed (Participants) | 21
  Without physical pain relieving measures during illumination | 8.1 (2.0)
  With physical pain relieving measures during illumination: number analyzed (Participants) | 79
  With physical pain relieving measures during illumination | 7.3 (2.2)

8. Primary Outcome: Changes in Blood Pressure (Systolic and Diastolic)
Description: Change from baseline is presented. The first measurement at Visit 2 (arrival at site) was considered as baseline value for all following measurements. Blood pressure was measured in mmHg. At Visit 2, photodynamic therapy was performed.
Time Frame: All visits through study completion after Visit 1: Visit 2, baseline, treatment day; Visit 3, approx. 7 days post treatment; Visit 4, approx.14 days post treatment; Visit 5, approx. 28 days post treatment
Population: One subject had elevated systolic and diastolic blood pressure at Visit 1 which was considered clinically significant and thus documented as relevant medical history. At Visit 2, blood pressure data was missing for one subject for the timepoint 'within 10 min prior to illumination', and for two subjects for the timepoint '60 min after illumination'. One subject missed Visit 3 and thus had no vital sign measurements at Visit 3.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
mmHg
  Systolic blood pressure - Visit 2 : Within 10 min before illumination: number analyzed (Participants) | 99
  Systolic blood pressure - Visit 2 : Within 10 min before illumination | 5.7 (12.8)
  Systolic blood pressure - Visit 2 : Within 10 min after illumination | 17.3 (16.5)
  Systolic blood pressure - Visit 2 : 60 min after illumination: number analyzed (Participants) | 98
  Systolic blood pressure - Visit 2 : 60 min after illumination | 10.8 (15.0)
  Systolic blood pressure - Visit 3: number analyzed (Participants) | 99
  Systolic blood pressure - Visit 3 | 1.1 (12.5)
  Systolic blood pressure - Visit 4 | -1.1 (13.4)
  Systolic blood pressure - Visit 5 | -0.9 (14.5)
  Diastolic blood pressure - Visit 2 : Within 10 min before illumination: number analyzed (Participants) | 99
  Diastolic blood pressure - Visit 2 : Within 10 min before illumination | 2.3 (6.6)
  Diastolic blood pressure - Visit 2 : Within 10 min after illumination | 7.1 (9.3)
  Diastolic blood pressure - Visit 2 : 60 min after illumination: number analyzed (Participants) | 98
  Diastolic blood pressure - Visit 2 : 60 min after illumination | 4.4 (7.9)
  Diastolic blood pressure - Visit 3: number analyzed (Participants) | 99
  Diastolic blood pressure - Visit 3 | 1.0 (8.8)
  Diastolic blood pressure - Visit 4 | -0.6 (8.3)
  Diastolic blood pressure - Visit 5 | 0.8 (8.5)

9. Primary Outcome: Changes in Pulse Rate
Description: Change from baseline is presented. The first measurement at Visit 2 (arrival at the site) was considered as baseline value for all following measurements. Pulse rate was measures in beats/min. At Visit 2, photodynamic therapy was performed.
Time Frame: as for outcome 8
Population: At Visit 2, pulse rate data was missing for one subject for the timepoint 'within 10 min prior to illumination', and for two subjects for the timepoint '60 min after illumination'. One subject missed Visit 3 and thus had no vital sign measurements at Visit 3.
Measure: Mean (Standard Deviation); unit: beats per min
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
beats per min
  Visit 2 : Within 10 min prior to illumination: number analyzed (Participants) | 99
  Visit 2 : Within 10 min prior to illumination | -2.1 (10.0)
  Visit 2 : Within 10 min after illumination | -1.2 (10.2)
  Visit 2 : 60 min after illumination: number analyzed (Participants) | 98
  Visit 2 : 60 min after illumination | -2.8 (9.5)
  Visit 3: number analyzed (Participants) | 99
  Visit 3 | 0.7 (9.8)
  Visit 4 | 0.7 (10.0)
  Visit 5 | 1.0 (9.2)

10. Primary Outcome: Changes in Body Temperature
Description: Change from baseline is presented. The first measurement at Visit 2 (arrival at site) was considered as baseline value for all following measurements. Body temperature was measured in °F and was converted to °C in the electronic Case Report Form. At Visit 2, photodynamic therapy was performed.
Time Frame: as for outcome 8
Population: At Visit 2, body temperature data was missing for one subject for the timepoint 'within 10 min prior to illumination', and for three subjects for the timepoint '60 min after illumination'. One subject missed Visit 3 and thus had no vital sign measurement at Visit 3. For one other subject, no temperature data was available at Visit 3.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
°C
  Visit 2 : Within 10 min prior to illumination: number analyzed (Participants) | 99
  Visit 2 : Within 10 min prior to illumination | -0.11 (0.41)
  Visit 2 : Within 10 min after illumination | -0.17 (0.60)
  Visit 2 : 60 min after illumination: number analyzed (Participants) | 97
  Visit 2 : 60 min after illumination | -0.08 (0.43)
  Visit 3: number analyzed (Participants) | 98
  Visit 3 | 0.04 (0.40)
  Visit 4 | -0.05 (0.39)
  Visit 5 | -0.03 (0.39)

11. Primary Outcome: Investigation of Clinical Chemistry Parameters
Description: Findings which differ from reference range and are considered to be clinically significant are to be reported. Clinical chemistry parameters include glucose, creatinine, total bilirubin, aspartate aminotransferase (AST), alanineaminotransferase (ALT), lactate dehydrogenase (LDH), alkalinephosphatase (AP),gamma glutamyl transferase (GGT), potassium, sodium, calcium, total protein, albumin.
Time Frame: At screening (Visit 1, up to 14 days before treatment) and at Visit 5 (approx. 28 days post treatment)
Population: Visit 1: For one subject, clinical chemistry but no hematology parameters were analyzed, as the sample arrived at the analyzing laboratory too late. However, no clinical chemistry measurements were documented for this subject. One other subject had no blood sample collected at Visit 1. Visit 5: One subject had no hematology and clinical chemistry assessment at Visit 5, as the blood sample was inadvertently not collected.
Measure: Number; unit: participants with findings considered CS
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
participants with findings considered CS
  Visit 1 (Overall): number analyzed (Participants) | 98
  Visit 1 (Overall) | 1
  Visit 1 - elevated blood glucose: number analyzed (Participants) | 98
  Visit 1 - elevated blood glucose | 1
  Visit 5 (Overall): number analyzed (Participants) | 99
  Visit 5 (Overall) | 2
  Visit 5 - elevated alanine aminotransferase: number analyzed (Participants) | 99
  Visit 5 - elevated alanine aminotransferase | 1
  Visit 5 - elevated aspartate aminotransferase: number analyzed (Participants) | 99
  Visit 5 - elevated aspartate aminotransferase | 1
  Visit 5 - elevated gamma glutamyl transferase: number analyzed (Participants) | 99
  Visit 5 - elevated gamma glutamyl transferase | 2
  Visit 5 - elevated blood glucose: number analyzed (Participants) | 99
  Visit 5 - elevated blood glucose | 1

12. Primary Outcome: Investigation of Hematology Parameters
Description: Findings which differ from reference range and are considered to be clinically significant are to be reported. Hematology parameters include hemoglobin, hematocrit, red blood cell count, leukocyte count (white blood cells(WBC)) with differential count (neutrophils, lymphocytes, monocytes, eosinophils, basophils), and platelet count.
Time Frame: At screening (Visit 1, up to 14 days before treatment) and at Visit 5 (approx. 28 days post treatment)
Population: as for outcome 11
Measure: Number; unit: participants with findings considered CS
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
participants with findings considered CS
  Visit 1: number analyzed (Participants) | 98
  Visit 1 | 0
  Visit 5: number analyzed (Participants) | 99
  Visit 5 | 0

13. Primary Outcome: Investigation of Urinalysis Parameters
Description: Findings which differ from reference range and are considered to be clinically significant (CS) are to be reported
Time Frame: At screening (Visit 1, up to 14 days before treatment) and at Visit 5 (approx. 28 days post treatment)
Population: Reasons for missing urinalysis data for 3 subjects at Visit 5 were "study coordinator error" (n=2) and "urinalysis inadvertently not collected" (n=1).
Measure: Number; unit: participants with findings considered CS
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
participants with findings considered CS
  Visit 1 | 0
  Visit 5: number analyzed (Participants) | 97
  Visit 5 | 0

14. Primary Outcome: Physical Examination of Head, Neck, Skin, Lymph Nodes, Thorax Including Heart and Lungs, Abdomen, and Musculoskeletal, Peripheral Vascular and Nervous System Status
Description: Abnormal findings, considered to be clinically significant (CS), are to be reported
Time Frame: At screening (Visit 1, up to 14 days before treatment) and at Visit 5 (approx. 28 days post treatment)
Population: At Visit 1, one participant had findings considered clinically significant. Of this 1 participant, these findings concerned the nervous system.
Measure: Number; unit: participants with findings considered CS
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
participants with findings considered CS
  Visit 1 | 1
  Of these: Findings concerning the nervous system: number analyzed (Participants) | 1
  Of these: Findings concerning the nervous system | 1
  Visit 5 | 0

15. Primary Outcome: Memory Tests
Description: Including picture- and question-based memory tasks; abnormal findings that are considered clinically significant will be documented
Time Frame: At screening (Visit 1, up to 14 days before treatment) and at Visit 2 (treatment day 1)
Population: Four subjects had missing data at Visit 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
Participants
  Visit 1 - All pictures memorized correctly: number analyzed (Participants) | 96
  Visit 1 - All pictures memorized correctly: No answer | 0
  Visit 1 - All pictures memorized correctly: Yes | 96
  Visit 1 - All pictures memorized correctly: No | 0
  Visit 1 - Questions on personal identification answered correctly: number analyzed (Participants) | 96
  Visit 1 - Questions on personal identification answered correctly: No answer | 0
  Visit 1 - Questions on personal identification answered correctly: Yes | 96
  Visit 1 - Questions on personal identification answered correctly: No | 0
  Visit 1 - Day of the week answered correctly: number analyzed (Participants) | 96
  Visit 1 - Day of the week answered correctly: No answer | 0
  Visit 1 - Day of the week answered correctly: Yes | 96
  Visit 1 - Day of the week answered correctly: No | 0
  Visit 1 - Arrival at site answered correctly: number analyzed (Participants) | 96
  Visit 1 - Arrival at site answered correctly: No answer | 2
  Visit 1 - Arrival at site answered correctly: Yes | 94
  Visit 1 - Arrival at site answered correctly: No | 0
  Visit 1 - 'Why here' answered correctly: number analyzed (Participants) | 96
  Visit 1 - 'Why here' answered correctly: No answer | 0
  Visit 1 - 'Why here' answered correctly: Yes | 96
  Visit 1 - 'Why here' answered correctly: No | 0
  Visit 2; prior PDT - All pictures memorized correctly: No answer | 0
  Visit 2; prior PDT - All pictures memorized correctly: Yes | 100
  Visit 2; prior PDT - All pictures memorized correctly: No | 0
  Visit 2; prior PDT - Questions on personal identification answered correctly: No answer | 0
  Visit 2; prior PDT - Questions on personal identification answered correctly: Yes | 100
  Visit 2; prior PDT - Questions on personal identification answered correctly: No | 0
  Visit 2; prior PDT - Day of the week answered correctly: No answer | 0
  Visit 2; prior PDT - Day of the week answered correctly: Yes | 99
  Visit 2; prior PDT - Day of the week answered correctly: No | 1
  Visit 2; prior PDT - Arrival at site answered correctly: No answer | 1
  Visit 2; prior PDT - Arrival at site answered correctly: Yes | 99
  Visit 2; prior PDT - Arrival at site answered correctly: No | 0
  Visit 2; prior PDT - 'Why here' answered correctly: No answer | 5
  Visit 2; prior PDT - 'Why here' answered correctly: Yes | 95
  Visit 2; prior PDT - 'Why here' answered correctly: No | 0
  Visit 2; after end of illumination - All pictures memorized correctly: No answer | 0
  Visit 2; after end of illumination - All pictures memorized correctly: Yes | 99
  Visit 2; after end of illumination - All pictures memorized correctly: No | 1
  Visit 2; after end of illumination - Questions on personal identification answered correctly: No answer | 0
  Visit 2; after end of illumination - Questions on personal identification answered correctly: Yes | 100
  Visit 2; after end of illumination - Questions on personal identification answered correctly: No | 0
  Visit 2; after end of illumination - Day of the week answered correctly: No answer | 0
  Visit 2; after end of illumination - Day of the week answered correctly: Yes | 100
  Visit 2; after end of illumination - Day of the week answered correctly: No | 0
  Visit 2; after end of illumination - Arrival at site answered correctly: No answer | 1
  Visit 2; after end of illumination - Arrival at site answered correctly: Yes | 99
  Visit 2; after end of illumination - Arrival at site answered correctly: No | 0
  Visit 2; after end of illumination - Remembered PDT: No answer | 14
  Visit 2; after end of illumination - Remembered PDT: Yes | 85
  Visit 2; after end of illumination - Remembered PDT: No | 1
  Visit 2; after end of illumination - 'Why here' answered correctly: No answer | 4
  Visit 2; after end of illumination - 'Why here' answered correctly: Yes | 96
  Visit 2; after end of illumination - 'Why here' answered correctly: No | 0

16. Primary Outcome: Neurological Investigations
Description: Including investigation of pupils (equality), coordination (finger-nose test), gait (balance), and sensitivity (cheeks, arms, legs); abnormal findings that are considered clinically significant (CS) will be documented
Time Frame: At screening (Visit 1, up to 14 days before treatment) and at Visit 2 (treatment day 1)
Population: One subject had no sensitivity assessment at Visit 1, and one other subject had no sensitivity assessment at Visit 2 after end of illumination.
Measure: Number; unit: participants with findings considered CS
Arm/Group | Total (BF-200 ALA)
Number analyzed (Participants) | 100
participants with findings considered CS
  Visit 1 - Pupils | 0
  Visit 1 - Coordination | 0
  Visit 1 - Gait | 0
  Visit 1 - Sensitivity: number analyzed (Participants) | 99
  Visit 1 - Sensitivity | 0
  Visit 2 prior PDT - Pupils | 0
  Visit 2 prior PDT - Coordination | 0
  Visit 2 prior PDT - Gait | 0
  Visit 2 prior PDT - Sensitivity | 0
  Visit 2 after end of illumination - Pupils | 0
  Visit 2 after end of illumination - Coordination | 0
  Visit 2 after end of illumination - Gait | 0
  Visit 2 after end of illumination - Sensitivity: number analyzed (Participants) | 99
  Visit 2 after end of illumination - Sensitivity | 0

ADVERSE EVENTS:
Time Frame: Collection of adverse events (AEs) starts with signing the informed consent (ICF (≤ 14 days prior to investigational medicinal product (IMP) application) documents until the final Visit (Visit 5, approx. 4 weeks after IMP application). For each subject the duration of the study was approx. 6 weeks (screening up to Visit 5).
Description: AEs will be discriminated as pre-treatment adverse events (PTAEs) and treatment emergent adverse events (TEAEs).
  AEs developing between signing the ICF (Visit 1) and investigational medicinal product (IMP) application at Visit 2 will be considered as PTAEs and documented as an AE. TEAEs are defined as all AEs or SAEs with onset or worsening after treatment with IMP at Visit 2 up to Visit 5.
Arm/Group | Total (BF-200 ALA)
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 100/100
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total (BF-200 ALA) (N=100)
Dry eye (Eye disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Application site discharge (General disorders) | 4 (4) — General disorders and administration site conditions
Application site discolouration (General disorders) | 6 (6) — General disorders and administration site conditions
Application site discomfort (General disorders) | 11 (13) — General disorders and administration site conditions
Application site dryness (General disorders) | 4 (4) — General disorders and administration site conditions
Application site erosion (General disorders) | 16 (18) — General disorders and administration site conditions
Application site erythema (General disorders) | 86 (97) — General disorders and administration site conditions
Application site exfoliation (General disorders) | 87 (117) — General disorders and administration site conditions
Application site haemorrhage (General disorders) | 10 (10) — General disorders and administration site conditions
Application site hyperaesthesia (General disorders) | 10 (10) — General disorders and administration site conditions
Application site induration (General disorders) | 18 (18) — General disorders and administration site conditions
Application site oedema (General disorders) | 35 (40) — General disorders and administration site conditions
Application site pain (General disorders) | 96 (193) — General disorders and administration site conditions
Application site papules (General disorders) | 2 (2) — General disorders and administration site conditions
Application site paraesthesia (General disorders) | 15 (17) — General disorders and administration site conditions
Application site pruritus (General disorders) | 65 (79) — General disorders and administration site conditions
Application site scab (General disorders) | 49 (58) — General disorders and administration site conditions
Application site swelling (General disorders) | 6 (8) — General disorders and administration site conditions
Application site vesicles (General disorders) | 14 (16) — General disorders and administration site conditions
Application site warmth (General disorders) | 17 (20) — General disorders and administration site conditions
Chills (General disorders) | 5 (6)
Fatigue (General disorders) | 6 (6)
Hypothermia (General disorders) | 4 (4)
Application site pustules (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Blood pressure increased (Investigations) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Headache (Nervous system disorders) | 22 (24)
Poor quality sleep (Psychiatric disorders) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 17 (31)
Hypertension (Vascular disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the Study and results shall not be published in any form without prior consent of Sponsor. All decisions on the timing and content of publications/ presentations will be coordinated by Sponsor. A draft of any manuscript, talks, abstracts, and all similar material shall be submitted to sponsor at least sixty (60) days before submission of the final form to any journal, scientific conference, symposium, or program review committee prior to publication or other release.

DOCUMENTS (2):
  • Study Protocol (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT05060237/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT05060237/SAP_001.pdf